CLINICAL TRIAL: NCT02785575
Title: The Impact of an Adjusted Calculation Model Regarding Heparin and Protamine Dosing on Bleeding and Transfusions After Cardiac Surgery Compared With Standard Dosing: A Randomized Single Blind Trial
Brief Title: Adjusted Calculation of Heparin and Protamin Dosing and Correlation With Postoperative Bleeding and Transfusions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jan van der Linden, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/2210
Record Dates: First submitted 2016-05-20; First posted 2016-05-30 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Cardiac Surgery; Bleeding; Transfusion; Protamine Sulfate; Heparin
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- HeProCalc (Active Comparator): This arm receives heparin and protamine doses according to the novel HeProCalc calculation model.
  Interventions: Other: HeProCalc algorithm
- Traditional calculations (No Intervention): This arm receives heparin and protamine doses according to the standard protocol (using calculations with body weight and ACT)

INTERVENTIONS:
Other: HeProCalc algorithm — Heparin and protamine dosage calculated by the algorithm HeProCalc
  Arms: HeProCalc

SUMMARY:
The study will compare a novel calculation model (HeProCalc AB) with a standard weight-based and activated clotting time adjusted calculation for the dosing of Heparin and protamine and assess the impact on postoperative bleeding and blood transfusions after cardiac surgery.

DETAILED DESCRIPTION:
During cardiac surgery with cardiopulmonary bypass (CPB), efficient anticoagulation is required in order to avoid microscopic clot formation or, in worst case, massive lift threatening thrombus formation. Heparin is by far the most common drug used to prevent blood from coagulating during CPB. Activated clotting time (ACT) is a point-of-care test of fibrin clotting time that has to be well prolonged to initiate safe CPB.

Following weaning from CPB, heparin is reversed by protamine. Administration of excess doses of protamine may have a deleterious effect on coagulation and contribute to postoperative bleeding with need of blood transfusions. In connection with CPB management, heparin and protamin doses are commonly calculated using body weight and ACT. However, a new Heparin-Protamin-Calculation computer program (HeProCalc) has been developed to provide patient titrated dosing of both heparin and protamin. However, any benefits regarding postoperative bleeding and transfusions has not been thoroughly investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery with the use of cardiopulmonary bypass
* Indication and planned use of heparin and protamine

Exclusion Criteria:

* Inability to leave informed consent or understanding the outline of the study
* Known coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative bleeding | 12 hours after chest closure
  According to UDPB severe or massive bleeding,

SECONDARY OUTCOMES:
Postoperative transfusions | 12 hours after chest closure
  12 hours after chest closure
Bleeding according to other validated definitions | 12 hours after chest closure
  PLATO major or life-threatening bleeding, BART massive bleeding, BARC CABG-related bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
On a group level in the planned publication. Upon request we will will share de-identified original data.

REFERENCES:
- [Background] Kjellberg G, Sartipy U, van der Linden J, Nissborg E, Lindvall G. An Adjusted Calculation Model Allows for Reduced Protamine Doses without Increasing Blood Loss in Cardiac Surgery. Thorac Cardiovasc Surg. 2016 Sep;64(6):487-93. doi: 10.1055/s-0035-1558649. Epub 2015 Aug 13. PMID 26270199